CLINICAL TRIAL: NCT05230667
Title: Comparison of the Effect of Combined Glenohumeral Joint and Subdeltoid Bursa Injection With Platelet-rich Plasma (PRP), Corticosteroid, and Normal Saline in Addition to Physical Therapy for Treatment of Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lin-Fen Hsieh, Principal Investigator, Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20211209R; NSTC 111-2314-B-341-002 - (Other Grant/Funding Number: National Science and Technology Council); 2024SKHADR037 (Other: Shin Kong Wu Ho-Su Memorial Hospital)
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Frozen Shoulder; Adhesive Capsulitis; Shoulder; Platelet-rich Plasma; Corticosteroid; Injection
Keywords: Frozen shoulder; adhesive capsulitis; shoulder; platelet-rich plasma; corticosteroid; injection
MeSH Terms: conditions — Bursitis | interventions — Adrenal Cortex Hormones; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRP injection (PRP group) and physical therapy (Active Comparator): Patients in the PRP group will receive both shoulder joint (GHJ) and SASD bursa injection for 2 times in 2-week interval. PRP will be prepared by taking 10ml venous blood which is then mixed with 2ml of thrombin and centrifuged in a specially designed tube at 3400 rotations per minute (rpm) for 15 minutes. About 2ml PRP and 3ml platelet poor plasma (PPP) will be extracted, then 4ml 1% xylocaine will be added to make 9ml injectate. 6ml injectate will be injected into the posterior GHJ with a 7 cm 23-gauge needle under ultrasound (US) guidance. Another 3ml injectate will be injected into the SASD bursa of the affected shoulder with a 3.8 cm 22-gauge needle under US guidance. Physical therapy will be conducted for 8 weeks.
  Interventions: Other: Corticosteroid injection (CS group); Other: Normal saline injection (NS group)
- Corticosteroid injection (CS group) and physical therapy (Active Comparator): Three ml triamcinolone (1ml= 10mg), 4ml 1% xylocain, and 2ml normal saline to make a 9ml injectate is injected into the affected shoulder (6ml to posterior GHJ and 3 ml to SASD bursa) for 2 times in 2-week interval. The techniques of injection are the same as those used in the PRP injection. Physical therapy will be conducted for 8 weeks.
  Interventions: Other: PRP injection (PRP group); Other: Normal saline injection (NS group)
- Normal saline injection (NS group) and physical therapy (Active Comparator): Four 4ml 1% xylocaine mixed with 5ml normal saline will be injected into the affected GHJ (6ml) and SASD bursa (3ml) for 2 times in 2-week interval . The techniques of injection are the same as those used in the PRP injection. Physical therapy will be conducted for 8 weeks.
  Interventions: Other: PRP injection (PRP group); Other: Corticosteroid injection (CS group)

INTERVENTIONS:
Other: PRP injection (PRP group) — Patients in the PRP group will receive both shoulder joint (GHJ) and SASD bursa injection for one time. PRP will be prepared by taking 10ml venous blood which is then mixed with 2ml of thrombin and centrifuged in a specially designed tube at 3400 rotations per minute (rpm) for 15 minutes. About 2ml PRP and 3ml platelet poor plasma (PPP) will be extracted, then 4ml 1% xylocaine will be added to make 9ml injectate. 6ml injectate will be injected into the posterior GHJ with a 7 cm 23-gauge needle under ultrasound (US) guidance. Another 3ml injectate will be injected into the SASD bursa of the affected shoulder with a 3.8 cm 22-gauge needle under US guidance.
  Arms: Corticosteroid injection (CS group) and physical therapy; Normal saline injection (NS group) and physical therapy
Other: Corticosteroid injection (CS group) — Three ml triamcinolone (1ml= 10mg), 4ml 1% xylocain, and 2ml normal saline to make a 9ml injectate is injected into the affected shoulder (6ml to posterior GHJ and 3 ml to SASD bursa). The techniques of injection are the same as those used in the PRP injection.
  Arms: Normal saline injection (NS group) and physical therapy; PRP injection (PRP group) and physical therapy
Other: Normal saline injection (NS group) — Four 4ml 1% xylocaine mixed with 5ml normal saline will be injected into the affected GHJ (6ml) and SASD bursa (3ml). The techniques of injection are the same as those used in the PRP injection.
  Arms: Corticosteroid injection (CS group) and physical therapy; PRP injection (PRP group) and physical therapy

SUMMARY:
Frozen shoulder, adhesive capsulitis, shoulder, platelet-rich plasma, corticosteroid, injection.

DETAILED DESCRIPTION:
This is a prospective assessor-blinded randomized controlled trial. We plan to enroll 90 participants with frozen shoulder from the outpatient clinic of the Department of Physical Medicine and Rehabilitation in our hospital. The study protocol and consent form have been approved by our ethics committee. After detailed explanation about the content of this study, participant is asked to sign an informed consent. The patients will be randomly divided into three groups: 1). PRP injection (PRP group); 2). Corticosteroid injection (CS group); 3). Normal saline injection (NS group). Randomization will be assigned according to a random number from a computer program by a statistician. The patients and the evaluator are unknown which group the patients are allocated, but the physician who performs joint injection knows which group the patients are assigned.

ELIGIBILITY:
Inclusion Criteria:

1. age between 20 to 80 years old;
2. shoulder pain for ≥ 1 month;
3. > 30% loss of passive range of motion (ROM) of the affected shoulder in external rotation and/or abduction, comparing with the sound side;
4. visual analog scale for pain on maximal passive external rotation or abduction > 4;
5. an empty or soft end feel on passive external rotation, or abduction and/or presence of night pain or rest pain;
6. showing willing to attend regular physical therapy programs for 8 weeks.

Exclusion Criteria:

1. severe systemic disorders including cancer, stroke, or cardiopulmonary diseases;
2. uncontrolled DM;
3. rotator cuff tear or calcification of the affected shoulder;
4. fracture, dislocation, or arthritis of the shoulder due to rheumatic disorders;
5. a hard end feel on passive external rotation or abduction of the affected shoulder;
6. a history of drug allergy to local anesthetics or corticosteroids;
7. receiving corticosteroid or hyaluronic acid joint or bursa injection of the affected shoulder during the preceding three months.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
The Shoulder Pain and Disability Index (SPADI) | Change between baseline and at 1 months, 2 months, 4 months, 6 months after the beginning of the treatment.
  The SPADI is a self-administered questionnaire that evaluate the pain and disability of shoulder diseases. It has 2 subclasses (pain and disability) that consists of 13 items. The pain domain has 5 items and the disabilities domain has 8 items. The SPADI score, which ranges between 0 (best score) and 100 (worst score), is calculated by averaging the scores from the 2 subclasses.

SECONDARY OUTCOMES:
The pain visual analog scale (VAS) | Change between baseline and at 1 months, 2 months, 4 months, 6 months after the beginning of the treatment.
  The pain VAS is obtained using a 100-mm-long horizontal line, with 0 mm on the left, indicating no pain, and 100 mm on the right, indicating very severe pain.22 The pain at rest is defined as rest pain, and pain on maximal abduction of the affected shoulder is defined as activity pain. The reliability of pain VAS is 0.94, but in the absence of a criterion standard for pain, criterion validity cannot be evaluated.
Range of motion（ROM） | Change between baseline and at 1 months, 2 months, 4 months, 6 months after the beginning of the treatment.
  All the 4 planes of ROM will be measured. It includes abduction in the frontal plane, forward flexion, internal rotation, and external rotation with the arm at 0° of abduction.
Shoulder Disability Questionnaire（SDQ） | Change between baseline and at 1 months, 2 months, 4 months, 6 months after the beginning of the treatment.
  The SDQ is a pain-related questionnaire that contains 16 items describing common situations that may induce symptoms in patients with shoulder disorders. The response options are "yes," "no," and "not applicable." The final score is calculated by dividing the number of positively scored items by the total number of applicable items and then multiplying this number by 100, which results in a final score ranging between 0 (no disability) and 100 (the worst possible condition).
The 36-item Short Form Health Survey（SF-36） | Change between baseline and at 1 months, 2 months, 4 months, 6 months after the beginning of the treatment.
  The SF-36 is a generic measure of quality of life and is composed of 8 subscales related to the following components: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each subscale generates a score from 0 to 100, and higher scores indicate better health.
Self-assessment of the treatment effect | Change between baseline and at 1 months, 2 months, 4 months, 6 months after the beginning of the treatment.
  Patient's evaluation of the treatment effect consists of the answer to one question: "Is the treatment effective?" scored on a Likert scale (very effective=5, effective=4, same=3, worse=2, much worse=1).

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan